CLINICAL TRIAL: NCT01505673
Title: Adding Liraglutide to High Dose Insulin: Breaking the Cycle
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ildiko Lingvay (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Ildiko Lingvay, Assistant Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIS-000235
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: Insulin; Glucagon-like peptide; Liraglutide; Beta-Cell; pancreatic steatosis; hepatic steatosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Insulin Resistance; Fatty Liver | interventions — Liraglutide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Active Comparator)
  Interventions: Drug: Liraglutide
- Saline injection (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Liraglutide — Liraglutdie 1.8mg injected subcutaneously from pen device once daily for 6-months
  Other Names: Victoza
  Arms: Liraglutide
Drug: Saline — Placebo injection of 1.8mg saline once daily for 6-months
  Arms: Saline injection

SUMMARY:
The purpose of this study is to evaluate whether the addition of liraglutide 1.8 mg/day to a high-dose insulin regimen (>1.8 units/kg/day) in patients with uncontrolled (HbA1c >7.5%) type 2 diabetes mellitus will improve blood sugar control.

It also evaluates the effect of liraglutide on liver and pancreatic fat content, explores the mechanism of blood sugar improvement by assessing weight and pancreatic hormone release, and assesses blood pressure, lipid profile, and liver function. Finally it will look at patient quality of life and safety.

DETAILED DESCRIPTION:
Type 2 diabetes is a progressive disease with incessant beta-cell dysfunction that often ultimately requires insulin treatment. Patients requiring high insulin dosages represent a particular treatment challenge and often have uncontrolled glycemia despite progressive dose increases and are especially prone to insulin related lipotoxicity and weight gain.

Glucagon-like peptide agonists (GLP-1) such as liraglutide have many actions that position them to break the vicious cycle in this population through the following mechanisms: (1) weight loss; (2) improved hepatic steatosis; (3) improved pancreatic steatosis; (4) decreased glucagon levels; (5) improved beta-cell function.

The purpose of the study is to demonstrate that liraglutide is both effective and safe when added to a high dose insulin treatment regimen. Liraglutide will improve glycemic control, weight, metabolic parameters, as well as patient satisfaction, with minimal adverse events. The study also proposes to study the mechanisms through which such improvements might occur, especially beta-cell function, glucagon levels, and hepatic and pancreatic fat content.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Insulin dose of >1.8 units/kg/day (represents total daily insulin dose, regardless of formulation, regimen, number of daily shots)
* HbA1c ≥ 7.5% and ≤ 11%
* Age ≥ 18
* Stable comorbidities on stable treatment regimens
* Stable dose of all oral hypoglycemics for ≥ 3 months prior to enrollment
* Ability to provide informed consent before any trial-related activities

Exclusion Criteria:

* Type 1 diabetes mellitus
* Any contraindication to the MRI procedure (metallic implants, severe claustrophobia, pregnancy, unable to lie still on a hard table for the duration of the procedure, weight above 400 lb - limit of the MRI table, magnet's inner circumference smaller than the largest body circumference)
* History of any pancreatic disease as it might interfere with the pancreatic TG measurement (i.e. pancreatitis, tumors, cysts, type 1 diabetes, any pancreatic surgery)
* End Stage Renal Disease on dialysis due to increased risk of hypoglycemia, and possible interference with accurate measurement of HbA1c
* Incretin therapy (any GLP-1 agonist or DPP-IV inhibitor)
* Unstable or decompensated comorbidities
* Personal or family history of medullary thyroid carcinoma or MEN-2 syndrome
* Severe gastroparesis
* Pregnancy, breast feeding, intention to become pregnant, or not using adequate contraceptive measures
* Organ transplant recipient or waiting list candidate
* Steroid use (current or potential use during the trial)
* Known/suspected allergy to trial medication, excipients, or related products
* Contraindications to study medications, worded specifically as stated in the product's prescribing information
* Non-English speaking volunteers since no interpreters are available and the safety of the volunteers could be jeopardized if adequate and reliable communication is not possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ildiko Lingvay, MD, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern, Dallas, Texas, United States

REFERENCES:
- [Derived] Vanderheiden A, Harrison L, Warshauer J, Li X, Adams-Huet B, Lingvay I. Effect of Adding Liraglutide vs Placebo to a High-Dose lnsulin Regimen in Patients With Type 2 Diabetes: A Randomized Clinical Trial. JAMA Intern Med. 2016 Jul 1;176(7):939-47. doi: 10.1001/jamainternmed.2016.1540. PMID 27273731
- [Derived] Vanderheiden A, Harrison LB, Warshauer JT, Adams-Huet B, Li X, Yuan Q, Hulsey K, Dimitrov I, Yokoo T, Jaster AW, Pinho DF, Pedrosa I, Lenkinski RE, Pop LM, Lingvay I. Mechanisms of Action of Liraglutide in Patients With Type 2 Diabetes Treated With High-Dose Insulin. J Clin Endocrinol Metab. 2016 Apr;101(4):1798-806. doi: 10.1210/jc.2015-3906. Epub 2016 Feb 24. PMID 26909799

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liraglutide | Saline Injection
Started | 35 | 36
Completed | 32 | 34
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Saline Injection | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 36 | 71
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (8.1) | 55.5 (6.6) | 54.2 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 12 | 14 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 34 | 66

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control Measured by HbA1c
Description: HbA1c (%)
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: Percent HbA1c
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
Percent HbA1c | 7.9 (1.1) | 8.9 (1.3)

2. Secondary Outcome: Pancreatic and Hepatic Triglyceride Content
Description: Liver Triglyceride and Pancreatic Triglyceride
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: Percent Triglyceride
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
Percent Triglyceride
  Liver Triglyceride | 12.3 (5.8) | 12.2 (7.8)
  Pancreatic Triglyceride | 12.53 (8.13) | 14.64 (9.25)

3. Secondary Outcome: Weight
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
Kilograms | 114 (21) | 117 (27)

4. Secondary Outcome: Beta-Cell Function
Description: Fasting Glucose as a Measure of Beta-Cell Function
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
mg/dL | 179 (75) | 197 (98)

5. Secondary Outcome: Glucagon
Description: Measured during mixed meal challenge test.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
pg/mL | 107.3 (44.5) | 93.8 (37.8)

6. Secondary Outcome: Total Daily Insulin Dose
Description: The 3 days average of the total daily dose of insulin used within 3 consecutive days prior office visit 6 month.
Time Frame: 6-months
Measure: Median (Inter-Quartile Range); unit: IU
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
IU | 200 [163 to 275] | 218 [160 to 260]

7. Secondary Outcome: Number of Daily Injections
Description: The 3 days average of the number of daily injections performed within 3 consecutive days prior office visit 6 month.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: number/day
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
number/day | 3.7 (1.4) | 3.8 (1.3)

8. Secondary Outcome: Blood Pressure
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
mmHg
  Systolic | 134 (18) | 135 (17)
  Diastolic | 80.5 (13.7) | 74.3 (9.7)

9. Secondary Outcome: Lipid Profile
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
mg/dL
  Total cholesterol | 154 (41) | 152 (42)
  LDL | 83.9 (37.2) | 76.3 (28.4)
  HDL | 36.6 (9.8) | 37.6 (9.9)

10. Secondary Outcome: Liver Function Blood Test
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
U/L
  ALT | 25.8 (13.5) | 36.0 (43.7)
  AST | 26.4 (17.6) | 32.1 (30.0)

11. Secondary Outcome: Hypoglycemic Events
Description: Reported as hypoglycemic events per month by patient as any blood glucose <70 mg/dl or symptoms of hypoglycemia with blood glucose >70 mg/dl
Time Frame: 6-months
Measure: Median (Inter-Quartile Range); unit: events per month per patient
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
events per month per patient | 1.1 [0.7 to 1.7] | 0.7 [0.5 to 1.2]

12. Secondary Outcome: Quality of Life Survey (QoL) - General Health Perception
Description: General health perception was measured at randomization and 6 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 1-5, where 1 = excellent; 2 = very good; 3 = good; 4 = fair; 5 = poor.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
score on a scale | 3.1 (0.9) | 3.6 (0.6)

13. Secondary Outcome: Beta-Cell Function
Description: Fasting C-peptide as a Measure of Beta-Cell Function
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: microgram/L
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
microgram/L | 2.48 (1.18) | 1.75 (1.19)

14. Secondary Outcome: Matsuda Index as a Measure of Beta Cell Function
Description: The Matsuda index is a measure of insulin sensitivity and has no minimum/maximum values. Index values are calculated as 500,000/square root of ((fasting glucose x fasting c-peptide x 333) x (mean 120 min post-meal glucose x mean 120 min post-meal c-peptide x 333)). Higher/lower values = better/worse insulin sensitivity.
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: index
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
index | 2.88 [1.67 to 3.70] | 3.12 [1.78 to 9.70]

15. Secondary Outcome: Beta-cell Function
Description: AUC c-peptide
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: ug/(L/min)
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
ug/(L/min) | 1234.6 (588.6) | 922.9 (470.5)

16. Secondary Outcome: Ratio (AUC C-peptide/AUC Glucose)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
Ratio | 0.019 (0.010) | 0.013 (0.008)

17. Secondary Outcome: AUC Glucose
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/(dL/min)
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
mg/(dL/min) | 71747 (22141) | 79278 (29416)

18. Secondary Outcome: Quality of Life Survey (QoL) - Current Health Perception
Description: Current health perception was measured at randomization and 6 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 1-5, where 1 = much better than 3 months ago; 2 - Somewhat better now than 3 months ago; 3 - About the same; 4 - Somewhat worse now than 3 months ago; 5 Much worse now than 3 months ago.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
score on a scale | 2.1 (0.9) | 2.6 (1.0)

19. Secondary Outcome: Quality of Life Survey (QoL) - Treatment Satisfaction
Description: Quality of Life Survey (QoL) - treatment satisfactionTreatment satisfaction was measured at randomization and 6 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 1-5, where 1 - very satisfied; 2 - moderately satisfied; 3 - neither satisfied nor dissatisfied; 4 - moderately dissatisfied; 5 - very dissatisfied.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
score on a scale | 2.4 (0.8) | 2.7 (0.7)

20. Secondary Outcome: Quality of Life Survey (QoL) - Treatment Impact
Description: Treatment impact was measured at randomization and 6 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 1-5, where 1 - very satisfied; 2 - moderately satisfied; 3 - neither satisfied nor dissatisfied; 4 - moderately dissatisfied; 5 - very dissatisfied.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
score on a scale | 2.3 (0.5) | 2.6 (0.7)

21. Secondary Outcome: Quality of Life Survey (QoL) - Social or Vocational Worry
Description: Social or vocational worry was measured at randomization and 6 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 0-5, where 0 - does not apply; 1 - never; 2 - seldom; 3 - sometimes; 4 - often; 5 - all of the time.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
score on a scale | 1.5 (0.7) | 1.0 (0.9)

22. Secondary Outcome: Quality of Life Survey (QoL) - Hypoglycemia Fear
Description: Hypoglycemia fear was measured at randomization and 6 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 1-5, where 1 - never worry; 2 - rarely water; 3 - sometimes worry; 4 - often worry; 5 - very often worry.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
score on a scale | 1.9 (0.7) | 2.0 (0.8)

23. Secondary Outcome: Quality of Life Survey (QoL) - Glycemia Control Perception
Description: Glycemia control perception was measured at randomization and 6 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a scale score of 1-7, where 1 - extremely controlled and 7 - not at all controlled.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
score on a scale | 2.0 (1.0) | 2.9 (1.0)

24. Secondary Outcome: Quality of Life Survey (QoL) - Lifestyle Flexibility
Description: Lifestyle flexibility was measured at randomization and 6 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 1 to 5, where 1 - a great deal of choice; 2 - a lot of choice; 3 - some choice; 4 - a little choice; 5 - no choice.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
score on a scale | 2.2 (0.9) | 2.6 (0.7)

25. Secondary Outcome: Quality of Life Survey (QoL) - Social Stigma
Description: Social stigma was measured at randomization and 6 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 1 to 5, where 1 strongly agree; 2 - somewhat agree; 3 - neither agree nor disagree; 4 - somewhat disagree; 5 - strongly disagree.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
score on a scale | 2.5 (1.1) | 2.4 (1.0)

26. Secondary Outcome: Quality of Life Survey (QoL) - Satisfaction With Insulin Treatment
Description: Satisfaction with insulin treatment was measured at randomization and 6 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a scale score of 1 to 7, where 1 extremely satisfied to 7 - not at all satisfied.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
score on a scale | 1.6 (1.0) | 2.3 (1.3)

27. Secondary Outcome: Quality of Life Survey (QoL) - Willingness to Continue Insulin Treatment
Description: Willingness to continue insulin treatment was measured at randomization and 6 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a scale score of 1 to 7, where 1 extremely willing to 7 - not at all willing.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liraglutide | Saline Injection
Number analyzed (Participants) | 32 | 34
score on a scale | 1.0 (0.5) | 2.1 (1.3)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Liraglutide: Liraglutide: Liraglutide 1.8mg injected subcutaneously from pen device once daily for 6-months
Arm/Group | Liraglutide | Saline Injection
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/35 | 6/36
Other Adverse Events (participants affected / at risk) | 14/35 | 14/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=35) | Saline Injection (N=36)
Atrial fibrilation (Cardiac disorders) | 1 (1) | 0 (0)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stent placement (Cardiac disorders) | 0 (0) | 2 (2)
Acute cholecystitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=35) | Saline Injection (N=36)
Nausea (Gastrointestinal disorders) | 11 (11) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Decreased in apetite (Gastrointestinal disorders) | 6 (6) | 4 (4)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Increase of serum amylase (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No